CLINICAL TRIAL: NCT04337554
Title: Exoskeleton Footwear to Improve Walking Performance and Subject-reported Preference
Brief Title: Exoskeleton Footwear to Improve Walking
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Nebraska (Other); Results Group LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: A3266-R
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Peripheral Arterial Disease
Keywords: Exoskeleton Device
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Older healthy: Individuals over 40 years of age
  Interventions: Device: Exoskeleton footwear
- Peripheral artery disease: Individuals over 40 years of age with peripheral artery disease.
  Interventions: Device: Exoskeleton footwear

INTERVENTIONS:
Device: Exoskeleton footwear — Assistive footwear

SUMMARY:
The purpose of this study is to determine the best assistance level of an exoskeleton footwear (EF) that can assist walking for people older than 40 with and without peripheral artery disease (PAD). The test will be performed on two different groups of people for this study that include: 1) people with PAD, and 2) individuals who don't have PAD.

Data will be collected from 50 healthy older individuals and 25 patients with PAD, both groups will be 40 years or older.

Gait biomechanics, muscle oxygenation, and energy cost for seven different walking conditions including normal walking, walking with EF with no assistance, and walking with EF with 5 different levels of assistance will be collected from the healthy older individuals. Additionally, subject-reported outcomes after each walking conditions including perceived comfort and fatigue, rate of perceived exertion and feasibility of the EF will be collected.

Gait biomechanics, muscle oxygenation, energy cost, and patient-reported outcomes will be measured in patients with PAD for four walking conditions including normal walking, walking with EF but no assistance, walking with EF with the best two assistance levels. Subjects will be allowed to acclimate to the EF prior to recording data. All patients with PAD will participate in feasibility interviews that will assess acceptability, demand, implementation, and practicality.

All subjects will be asked to fill out questionnaires that assess quality of life, physical function, and the ability to complete activities of daily living.

DETAILED DESCRIPTION:
Claudication due to peripheral artery disease (PAD) causes patients to walk less and slower, lose independence in daily living activities, and be sedentary compared to their healthy counterparts. The investigators' research has identified functional limitations in the walking patterns of claudicating patients. The most prominent and consistent deficit is of the posterior calf muscles, the ankle plantarflexors, to generate healthy ankle torque and power during walking. Previous work in the investigators' laboratory has established that these functional deficits are related to the presence of a myopathy in the legs of patients with PAD which is characterized by myofiber degeneration and muscle fibrosis. An intervention that compensates for impaired muscle physiology and performance is needed to improve walking ability and independence in patients with PAD.

The long-term goal of this project is to improve the quality of life of patients with PAD by using assistive exoskeletons. Currently, there is a critical treatment gap for those patients with PAD whose disease presentation does not warrant operative revascularization (based on risk-benefit analysis that considers multiple factors including disease severity, comorbid conditions and operative risk), but who desire to regain their walking ability and independence. Ankle-foot orthoses have recently been implemented to reduce the demands for biological ankle plantarflexor torque and to compensate for power deficiency. Biological ankle torque/power is torque/power generated by the plantarflexor muscles apart from that provided by an assistive device. The investigators have developed a lightweight and low-cost 3D printable elastic exoskeleton and footwear combination called exoskeleton footwear (EF). The EF assists with push-off by using springs that mimic ankle plantarflexor forces. Exoskeletons that assist propulsion address both the myopathy and low blood flow problems associated with claudication. Mechanical force from the EF compensates for insufficient muscle propulsion force, while decreasing blood flow demand and the muscular stress caused by ischemia. A properly designed exoskeleton will likely allow patients with PAD to walk longer without pain or walk the distance needed for completing daily activities with less stress to the affected leg. As a first step the investigators propose to determine the effect of EF on walking performance, focusing on how different levels of EF support contribute to changes in the biological ankle torque and power, energy cost, and calf muscle oxygenation. The investigators will test healthy older adults to ensure and confirm comfort, low risk of injury to the foot and calf, and high potential for device adoption in patients with PAD.

The EF will then be evaluated in patients with PAD. Healthy older individuals are selected for the initial phase of the project because, like patients with PAD, they produce less push-off torque and power during walking compared with healthy young; making them an appropriate model for PAD limitations. Furthermore, compared to patients with PAD, healthy older can tolerate longer walking trials, which are necessary to identify effective device parameters and also have a significantly lower risk of developing foot and calf injuries while the comfort and shape of the EF are assessed and adjusted to accommodate individuals with different foot and leg morphologies.

Hypothesis: Walking performance will improve with EF in healthy older and patients with PAD. The investigators hypothesize there will be an EF assistance level to satisfy subject-reported preference and walking performance goals.

Specific Aim 1: To determine the levels of EF assistance force which produce better walking performance in older subjects. Improvements in walking performance will be assessed by measuring how different levels of EF assistance contribute to changes in the biological ankle torque and power during push-off, the energy cost of walking, and the calf muscle oxygenation during walking.

Specific Aim 2: To determine the levels of EF assistance force which produce better subject-reported preference in older subjects. Preference will be measured using visual-analog scales, perceived exertion and pain questionnaires, and interview-style surveys about acceptability (satisfaction, intent to use), demand (perceived demand), and practicality (effects, ability of participants to use EF).

Specific Aim 3: To determine the effect of EF assistance levels on walking performance and subject-reported preference in patients with PAD. Results from Aims 1 and 2 will guide the assistance levels tested in this aim.

Research Design and Methods Healthy elderly will be evaluated in a total of seven conditions in Aims #1 and #2: five different EF stiffness levels including EF: Stiffness 1 (5.6 kN/m), EF Stiffness 2 (7.9 kN/m), EF Stiffness 3 (10.5 kN/m), EF Stiffness 4 (13.3 kN/m), EF Stiffness 5 (17.2 kN/m), EF with a disengaged spring and one normal walking condition (no EF).

PAD patients will be evaluated in four conditions in Aim #3: two different EF stiffness levels, one condition in which the subjects will wear the EF with a disengaged spring and one normal walking condition (no EF). Spring stiffness will be adjusted as a function of body mass to provide a normalized torque input across subjects. These stiffness levels were chosen based on previous research work using a similar, device in healthy young individuals. The EF will be set to release the spring at 42% of the stride. Increases in energy cost at stiffness values above and below the optimal value will be an indicator the stiffness levels are within the appropriate scale. Healthy older adults and patients with PAD will be tested to determine the effect of EF assistance force on walking performance and energy cost and subject-reported preference with varying EF assistance levels

A total of 50 adults, ages 50 years and older from the Nebraska and Western Iowa Veterans Affairs' Medical Center (VAMC) and the surrounding Omaha community to complete Aims 1 and 2 will be recruited. Aim 3 will include 25 patients with PAD recruited from the VAMC.

Data collection Protocol for Aims #1 and #2:

Walking: Subjects will complete seven minutes of walking at their preferred walking speed on an instrumented treadmill (AMTI, Watertown, MA) while kinetics and kinematics are captured at 100 Hz with a 17 camera digital motion capture system (Cortex 6.2, Motion Analysis Corp, Santa Rosa, CA). The three minutes of walking will be for subjects to get accustomed to the new assistance level in the EF. Preferred walking speed will be determined prior to collecting any data and it will be held consistent across the seven conditions.

Subject will also walk on flat ground for seven different conditions.

Muscle Oxygenation: Bilateral gastrocnemius muscle oxygenation (StO2) will be measured using continuous-wave near infrared spectroscopy (PortaMon, Artinis Medical System, Netherlands) before, during and after each treadmill walking condition (described above).

Energy cost: A portable metabolic cart will be used to measure gas exchange on a breath-by-breath basis, providing a measure of oxygen consumption during each of the seven treadmill walking conditions.

Perceived comfort and fatigue: A visual analog scale will be used to capture subjects' perception of comfort and fatigue after each treadmill and flat ground condition. The visual analog scale will range from 0 (low comfort; high fatigue) to 10 (high comfort; low fatigue).

Rate of perceived exertion: Self-reported perceived exertion values from the Borg Rate of Perceived Exertion scale (6 (no exertion) to 20 (maximal exertion)) will be recorded after each condition.

Data collection Protocol for Aims #3:

Walking performance and subject-reported preference will be assessed in the same manner as in Aims 1 and 2 except the treadmill walking test will be replaced with maximum walking distance tests (see description below). For this reason, testing will be divided into two days, with two maximum walking distances tests completed on each day. Subjects will rest until any claudication pain subsides between each maximum walking distance tests. Subjects will complete testing of the same outcomes (1-7 below) exactly as described in Aims 1 and 2 and maximum walking times (8 below). Maximum walking times are the best indicator of the implications of PAD on daily walking ability and participation in community activities.

All outcomes from the older subject's protocol will be assessed for PAD patients including 1) walking: On the treadmill test, biomechanics variables during the zero degree incline portion of the test will be collected. Rest time will be given between the conditions as needed for claudication pain to subside.

2) Muscle oxygenation, 3) Energy cost, 4) Perceived comfort and fatigue, 5) Rate of perceived exertion, 6) Feasibility.

Two additional outcomes measured for the PAD patients will be:

Perceived pain: Following the approach of perceived comfort and fatigue, a visual analog scale will be used to capture subjects' perception of pain after each condition. The visual analog scale will range from 0 (no pain) to 10 (intense pain) and will be assess after each EF condition.

Claudication Onset and Peak Walking Times: Walking ability will be determined with a progressive-load treadmill test with initial and maximum claudication distances as outcomes. Patients will walk on a treadmill that starts at 0% grade and 2.0 mph. Every two minutes, the grade will be increase by 2% up to a maximum of 15% grade, and the speed held constant throughout the test. The initial distance walked prior to the onset of pain (Claudication Onset Time - COT) and the distance patients walked until the test had to be stopped due to pain (Peak Walking Time -PWT) will be the outcome measures.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy older: At entry into the study, all subjects must:

* Be able to give written, informed consent
* Have a stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks as determined by a health history questionnaire
* Be 40 years of age or older

  * Healthy aged selected to match the population of patients with PAD
* Demonstrate negative history of chronic claudication or other exercise limitation as determined by a health history questionnaire

Inclusion criteria for patients with PAD: At entry into the study, all subjects must:

* Meet criteria 1-3 from above
* Demonstrate positive history of chronic claudication pain
* Demonstrate exercise-limiting claudication per history and direct observation
* Have evidence of occlusive disease on ankle/brachial index testing and/or computerized tomographic angiography

Exclusion Criteria:

Exclusion criteria for healthy older, any potential subjects will be excluded if they have:

* An ankle-brachial index < 0.90 at rest, as measured by the study team

  * Healthy subjects only
* Individuals without symptoms but with reduce blood flow (asymptomatic PAD) will be excluded
* Walking capacity limited by conditions affecting the legs (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Omaha VA Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
biological ankle torque in Newton meters/kilogram | baseline assessment
  The primary outcome variables of biological contribution to ankle torque and power will be calculated from five steps per leg during the flat ground walking. Ground reaction forces for the vertical, anterior-posterior, and medial-lateral direction, and joint angles, joint angular velocity for the hip, knee, and ankle during the stance phase of walking, joint torques and powers are will also be calculated.

SECONDARY OUTCOMES:
Muscle Oxygenation | baseline assessment
  Resting StO2, minimum StO2 during each treadmill trial, time to minimum StO2, and the StO2 recovery time will be calculated.
Energy cost | baseline assessment
  Steady-state oxygen consumption in ml/kg/min will be calculated from the final three minutes of the treadmill walking test.
Rate of perceived exertion | baseline assessment
  Self-reported perceived exertion values from the Borg Rate of Perceived Exertion scale (6 (no exertion) to 20 (maximal exertion)) will be recorded after each condition.
Claudication Onset and Peak Walking Times (seconds) | baseline assessment
  Subjects will perform a progressive-load treadmill test. During the treadmill test, patients will walk on a treadmill that starts at 0% grade and 2.0 miles/hour. Every two minutes, the grade will be increased by 2% up to a maximum of 15% grade and the speed will be held constant. Subjects will report claudication pain during the test. The initial distance walked prior to the onset of pain (Claudication Onset Time - COT) and the distance patients walked until the test had to be stopped due to pain (Peak Walking Time -PWT) will be the outcome measures.

CONTACTS AND LOCATIONS:
Overall Officials: Sara A. Myers, PhD, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE; Iraklis I Pipinos, MD, Principal Investigator — Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE
Locations (1):
- Omaha VA Nebraska-Western Iowa Health Care System, Omaha, NE, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-01-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT04337554/ICF_000.pdf